CLINICAL TRIAL: NCT00024804
Title: A Natural History Study of Bone and Mineral Disorders
Status: Recruiting | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010184; 01-D-0184
Record Dates: First submitted 2001-09-28; First posted 2001-10-01 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-12-04

CONDITIONS: Tumor Induced Osteomalcia; Osteomalacia; Familial Tumoral Calcinosis
Keywords: Natural History; skeletal diseases; Osteoporosis; Dysplasia; Osteomalacia; Bone Diseases; Skeletal Disease
MeSH Terms: conditions — Osteomalacia; Osteoporosis; Bone Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Subjects with known or suspected bone disease and disorder of mineral metabolism.

SUMMARY:
This study has four objectives: 1) to provide investigators the opportunity to study bone specimens from patients with various skeletal diseases; 2) to treat patients with skeletal diseases at the NIH; 3) to expose NIH trainees to certain skeletal diseases; and 4) to gain more knowledge about skeletal diseases and stimulate further study of bone biology.

Anyone with a disease that affects the skeleton may be eligible for this study.

All evaluations, tests, procedures and treatments given study participants are used in the standard care of skeletal diseases. No experimental evaluations or treatments are offered. Patient evaluations include a medical history, review of medical records and routine physical examination. Based on the findings, other procedures may be recommended, including blood tests, urine tests, and imaging tests, such as X-rays, bone densitometry, bone scan, computed tomography (CT) and magnetic resonance imaging (MRI).

Bone specimens from participants will be collected for research use. Specimens will be obtained from bone removed during a patient s planned surgical procedure performed for medical care, or patients may be requested to have a bone biopsy removal of a small piece of bone tissue as part of the patient evaluation procedure.

DETAILED DESCRIPTION:
Study Description:

To evaluate participants with bone and mineral disorders at the NIH Clinical Center and obtain tissue and clinical specimens from outside institutions

Objectives:

Primary Objective:

Provide a protocol within which participants with common and rare disorders of bone and mineral metabolism can be studied, evaluated and treated at NIH.

Secondary Objectives:

To obtain tissue and clinical specimens (including but not limited to blood, urine, nucleic acids, skin and bone) and data collected at outside institutions and the NIH Clinical Center from participants with various bone and mineral disorders.

Tertiary/Exploratory Objective:

Generate a pool of participants with bone and mineral disorders, from which research questions could arise and future clinical research studies may be generated.

Endpoints:

Primary Endpoint:

Medical evaluation with clinical assessments performed at time points specific to each participant s diagnosis. Analysis of research and participant outcome data will be performed.

Secondary Endpoint:

Genetic and/or biochemical assessments of surgical waste material from the NIH Clinical Center or other medical facilities.

Tertiary/Exploratory Endpoint:

Development of a database containing information from enrolled participants with bone and mineral disorders and annotated specimens and data.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population will include participants with known or suspected bone disease and/or with a known or suspected disorder of mineral metabolism. To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age 1 day of life or older
2. Have a known or suspected bone disease, as demonstrated by any one of the following: a fracture, or abnormal bone findings on x-ray, CT scan, MRI, or bone densitometry, and/or a medical or family history consistent with or suggestive of a bone disease.
3. Have a known or suspected disorder of mineral metabolism, as demonstrated by any one of the following: laboratory measurement above or below the reference values for either blood or urine calcium, phosphorus, magnesium, parathyroid hormone or vitamin D, or other measures of mineral metabolism, and/or a medical or family history consistent with or suggestive of a disorder of mineral metabolism.

EXCLUSION CRITERIA:

1. Participants unwilling or unable to abide by procedures of protocol.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with known or suspected bone disease and disorder of mineral metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-11-19 (Actual)

PRIMARY OUTCOMES:
Collection of clinical and research specimens | 10 years
  Specimens will be collected for creating better understanding of the disorders seen and for generating future research studies.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly B Roszko, M.D., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
As this study enrolls participants with a myriad of disorders and research specimens are not collected in a systematic manner, sharing of IPD is not meaningful.

REFERENCES:
- [Derived] Theng EH, Brewer CC, Oheim R, Zalewski CK, King KA, Delsmann MM, Rolvien T, Gafni RI, Braddock DT, Jeffrey Kim H, Ferreira CR. Characterization of hearing-impairment in Generalized Arterial Calcification of Infancy (GACI). Orphanet J Rare Dis. 2022 Jul 19;17(1):273. doi: 10.1186/s13023-022-02410-w. PMID 35854274
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-D-0184.html